CLINICAL TRIAL: NCT05609669
Title: Continuous And Data-drivEN CarE (CADENCE)
Brief Title: Continuous And Data-drivEN CarE (CADENCE) Pilot
Acronym: CADENCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY004953
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Related; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CADENCE program pilot (Experimental)
  Interventions: Other: CADENCE program

INTERVENTIONS:
Other: CADENCE program — The CADENCE program will consist of an integrated care pathway between the OBOT clinic, obstetric clinic, pediatric clinic, and behavioral health with multiple entry points, including emergency rooms, existing mobile harm reduction clinics, obstetric clinics, and delivery facilities. We also seek to provide wrap-around care for these families with peer support, care navigation, and robust community support, using existing Hillsborough County resources such as doula programs, Healthy Start, and other home visiting programs.

SUMMARY:
The proposed project seeks to use public health and clinical data on opioid use disorders (OUD) outcomes for mother and infants, which is the leading cause of death to mothers one year after deliver and can lead to neonatal withdrawal syndrome (NOWS) and other poor outcomes. Insufficient or incomplete data about OUD and lack of integrated programs for OUD treatment during pregnancy can be barriers to providing optimal care to mothers and infants.

DETAILED DESCRIPTION:
Maternal opioid use disorder (OUD) is the leading cause of maternal mortality in the first year after delivery nationwide. OUD also contributes substantially to out-of-home placements in the child welfare system. Medication for OUD (MOUD) is the primary standard of treatment, however, access to MOUD and prenatal care is limited, siloed, and fragmented in Florida. Gaps in access to and continuity of healthcare (prenatal, postpartum, pediatric, pharmacological and behavioral health) and other services for mothers in OUD recovery lead to poor outcomes for parent, child and family. There is also insufficient data integration, due to inconsistent data collection methods or use of diagnostic codes, to identify mother-infant dyads affected by OUD that could inform optimal care at the local level. Single-site studies that integrate substance use disorder programs in pregnancy have been shown to improve neonatal and maternal outcomes. With that in mind, the long-term goal of this study is to leverage high-quality local and timely data to improve OUD outcomes before, during, and after pregnancy with an integrated care approach that can be replicated throughout the state. The objective of the proposed project is to consolidate multiple streams of public health and clinical healthcare data to analyze equitable access and outcomes for families affected by maternal OUD for use in quality improvement cycles to rapidly refine our integrated CADENCE (Continuous and Data-Driven Care) Program. Our central hypothesis is that integrated, continuous, data-driven care will improve CADENCE patient outcomes. We will test this hypothesis through the following aims: 1) create an interactive data dashboard for maternal, neonatal, and infant outcomes for pregnancies affected by OUD; 2) pilot the CADENCE program and rapidly refine using a data-driven approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known opioid use disorder over the age of 18 years old who are pregnant

Exclusion Criteria:

* Patients without opioid use disorder, less than 18 years old, incarcerated, or non-pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
MOUD at delivery hospitalization | At delivery hospitalization
  Patients on subutex or methadone treatment at delivery hospitalization (yes/no)
Decreased pharmacologically treated NOWS | At delivery
  Medication clinically required for NOWS (yes/no)

SECONDARY OUTCOMES:
First trimester entry to prenatal care | Prenatal care, up to 40 weeks
  First prenatal care visit before 14 weeks gestational age (yes/no)
Prenatal care adequacy | Prenatal care, up to 40 weeks
  Kotelchuck index (score)
Hepatitis C screening | Prenatal care, up to 40 weeks
  Hepatitis C antibody screen collected during prenatal care (yes/no)
NICU admissions | At delivery hospitalization
  Admission to the NICU during delivery admission for any reason (yes/no)
Hospital length of stay (neonate) | At delivery hospitalization
  Number of days in hospital during delivery admission (#)
Department of Children and Families out-of-home placement | At delivery hospitalization
  Neonate placed in care of another family or with a foster family who is not the biological parents. This does not include planned adoptions. (yes/no)
Breastfeeding at discharge | At delivery hospitalization
  Exclusive breastfeeding at discharge from delivery admission (yes/no)
Enrollment in community supports and services. | Prenatal up to 1 year old
  Proportion of referrals to connection/enrollment in services (%)

OTHER OUTCOMES:
Acceptability of CADENCE Program | Prenatal up to 1 year old
  Patient satisfaction gauged by qualitative interview and quantitative surveys
Feasibility of CADENCE Program | Prenatal up to 1 year old
  Number of patients recruited per month, number of patients enrolled in program
Trialability of CADENCE Program | Prenatal up to 1 year old
  Ability to integrate into clinical flow as gauged by Clinical staff qualitative interview and quantitative surveys

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Marshall, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida/Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data: The raw data at the individual level will be available to users only under a specific data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. All data-sharing agreements must be approved by our institutional IRB and follow university protocols.
Access Criteria: Qualitative Data: The proposed research will include data from approximately 20 subjects. We will make the quantitative data, summary of qualitative data with representative quotes, and associated documentation available to users only under a specific data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Aggregate data and summary tables will be available through the NIH HEAL Initiative central data repository.